CLINICAL TRIAL: NCT01335087
Title: Impact of Sleep Apnea Syndrome in the Evolution of Acute Coronary Syndrome. Effect of Intervention With Continuous Positive Airway Pressure (CPAP). A Prospective Randomized Study. ISAACC Study
Brief Title: Continuous Positive Airway Pressure (CPAP) in Patients With Acute Coronary Syndrome and Obstructive Sleep Apnea (OSA)
Acronym: ISAACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: ResMed (Industry); Fondo de Investigacion Sanitaria (Other); EsteveTeijin Healthcare (Other); Spanish Society of Cardiology (Other); Sociedad Madrileña de Neumologia (Unknown)
Responsible Party: Principal Investigator, Ferran Barbe, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI10/02763
Record Dates: First submitted 2011-04-05; First posted 2011-04-14 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndrome; Obstructive Sleep Apnea
Keywords: sleep apnea; secondary prevention; cardiovascular endpoint
MeSH Terms: conditions — Acute Coronary Syndrome; Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Standard of Care; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lifestyle (Active Comparator): Standard care for OSA: lifestyle, and sleep hygiene counselling
  Interventions: Other: Standard care
- Continuous positive airway pressure CPAP (Experimental): CPAP treatment every night plus standard care for OSA: lifestyle, and sleep hygiene counselling
  Interventions: Other: Standard care; Device: continuous positive airway pressure
- Reference (No Intervention): This group will be followed according to cardiovascular protocols and will be evaluated as a reference group.

INTERVENTIONS:
Other: Standard care — Patients with conservative treatment: (Group 2). This group will also be instructed in hygienic-dietary measures, standard care of cardiovascular risk factors and sleep hygiene counselling.
  Arms: Continuous positive airway pressure CPAP; Lifestyle
Device: continuous positive airway pressure — Patients with CPAP treatment (Group 1): CPAP pressure titration will be performed by automated equipment before discharge. It will follow the methodology described by our group (Mass et al. Alternative Methods of titrating continuous positive airway pressure: a large multicentre study. American Journal of Respiratory and Critical Care Medicine (2004) vol. 170 (11) pp. 1218-1224). This group will also be instructed in hygienic-dietary measures recommended for all patients, standard care of cardiovascular risk factors and sleep hygiene counselling.
  Arms: Continuous positive airway pressure CPAP

SUMMARY:
OSA may be a modifiable risk factor for cardiovascular disease due to its association with hypertension, stroke, heart attack and sudden death. The standard therapy for symptomatic OSA is continuous positive airway pressure (CPAP). CPAP has been shown to effectively reduce snoring, obstructive episodes and daytime sleepiness and to modestly reduce blood pressure and other risk factors for cardiovascular disease. The overall aim of ISAACC is to determine if CPAP can reduce the risk of heart attack, stroke or heart failure for people with OSA admitted in a hospital for an acute coronary syndrome.

Overall objective:

To assess the impact of obstructive sleep apnea (OSA) and its treatment on the clinical evolution of patients with acute coronary syndrome (ACS).

Primary objectives:

1. To determine if continuous positive airway pressure (CPAP) treatment will reduce the rate of cardiovascular events (cardiovascular (CV) death, non-fatal events (acute myocardial infarction (AMI), non-fatal stroke, hospital admission for heart failure, and new hospitalizations) for unstable angina or transient ischaemic attack (TIA)) in patients with ACS and co-occurring sleep apnea.

Secondary objectives:

1. Determine the prevalence of OSA in patients who have suffered an episode of ACS.
2. Other secondary objectives will include the effects of CPAP on:

   * To evaluate a composite of CV death, myocardial infarction (MI) and ischaemic stroke.
   * Components of primary composite endpoints
   * Re-vascularization procedures
   * To evaluate all-cause death
   * To evaluate new onset, ECG-confirmed atrial fibrillation or other arrhythmias
   * To evaluate newly diagnosed diabetes mellitus, according to standard definitions
   * To evaluate OSA symptoms (Epworth Sleepiness Scale (ESS))
   * To evaluate quality of life in patients with ACS (Test EuroQol (EQ-5D).
3. To establish the relationship between the severity and phenotype of patients with OSA and clinical outcomes of ACS.
4. To establish the relationship between CPAP compliance and CV events incidence.
5. To identify biological risk markers that allow us to establish the most important mechanisms involved in cardiovascular complications in these patients.
6. To conduct a cost-effectiveness analysis of the diagnosis and CPAP treatment of patients with ACS who have obstructive sleep apnea.

DETAILED DESCRIPTION:
Methods:

Study design: multi-centre, open label, parallel, prospective, randomised, controlled trial.

Patients: We will include consecutive patients with an ACS diagnosis evaluated in participating Coronary Care Unit.

Study sites: IRB Lleida (Lleida), Hospital Son Dureta (Palma de Mallorca), Hospital Clínic (Barcelona), Hospital Germans Tries i Pujol (Barcelona), Hospital de Bellvitge (Barcelona), Hospital Sant Pau (Barcelona), Hospital Txagorritxu (Vitoria), Hospital de Cruces (Bilbao), Hospital San Pedro de Alcántara (Cáceres), Hospital Parc Taulí (Barcelona) and Hospital de Guadalajara (Guadalajara), Hospital de Vallecas (Madrid), Hospital de Yagüe (Burgos), Hospital de Requena (Valencia), Hospital San Juan, (Alicante), Hospital Central de Asturias (Oviedo).

Duration of the study: 3 years. Methodology: During a hospital stay we will assess the degree of daytime sleepiness (Epworth Scale) in patients treated at the Coronary Care Unit with a diagnosis of ACS. The results of this evaluation will define the inclusion of the patient in the study.

Patients with and ESS score ≤ 10 will be included in the study and will undergo a cardio-respiratory polygraphy. Patients with an AHI ≥ 15 h-1 will be randomized to CPAP treatment or conservative. Patients with and AHÍ < 15 h-1 will be followed as standard management according to cardiovascular protocols and will be evaluated as a reference group. Therefore, the study will have three groups, with a total of 1,864 patients, as follows: patients with an AHI ≥ 15 h-1 will be randomized to CPAP treatment (Group 1) (n=632) or conservative treatment (Group 2) (n=632). Patients with an AHI < 15 h-1 that will be followed as a reference group (Group 3) (n=600).

Patients with an ESS score higher than 10 will be excluded of the study and referred to the sleep unit of each participating center for evaluation.

Patients included in the study will be monitored and followed for a minimum of one year and a maximum of three years. Patients will be examined at the time of inclusion (T0), after one month (T1), three months (T2), six months (T3), 12 months (T4) and every six months thereafter, if applicable, during the follow-up period. Evaluations will include; i)new episodes of ACS, stroke, TIA, heart failure, hospitalization for cardiovascular causes and cardiovascular mortality, ii) biological risk markers involved in cardiovascular complications, iii) an evaluation of the cost-effectiveness of diagnosis and CPAP treatment in patients with ACS who have obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years old.
2. Patients admitted for documented symptoms of ACS with or without T segment elevation and have an hospital stay between 24h and 72 h in the moment to perform polygraphy .
3. Patients with and Epworth Sleep Scale score ≤ 10 (patients without excessive daytime sleepiness).
4. Written informed consent signed.

Exclusion Criteria:

1. Previous CPAP treatment for OSA diagnosis
2. Psycho-physical inability to complete questionnaires.
3. Presence of any previously diagnosed sleep disorders: narcolepsy, insomnia, chronic sleep deprivation, regular use of hypnotic or sedative medications and restless leg syndrome
4. Patients with > 50% of central apneas or the presence of Cheyne-Stokes Respiration (CSResp)
5. Patients with chronic diseases: neoplasia, renal failure (GFR<30 ml/min), severe chronic obstructive pulmonary disease, chronic depression and other very limiting chronic diseases.
6. A medical history that may interfere with the study objectives or, in the opinion of the investigator, compromise the conclusions.
7. Any medical factor, social or geographical, that may jeopardize patient compliance.(e.g., alcohol consumption (more 80 gr/day in men and more than 60 gr / day in women), no fixed address, disorientation, or a history of non-compliance).
8. Any process, cardiovascular or otherwise, that limits life expectancy to less than one year.
9. Patients in cardiogenic shock who have poor expectations for short-term outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1864 (Actual)
Dates: Start 2011-04; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Rate of cardiovascular events in patients with acute coronary syndrome and co-occurring sleep apnea. | 12 month after the inclusion of the last patient
  Cardiovascular events are: cardiovascular death, non-fatal AMI, non-fatal stroke, hospital admission for heart failure, and new hospitalization for unstable angina or TIA.

SECONDARY OUTCOMES:
Prevalence of OSA in patients who have suffered an episode of ACS. | 24 month (inclusion period)
  Determined at the inclusion of the patient
Composite of major CV events | 12 month after the inclusion of the last patient
  CV death, myocardial infarction (MI) and ischaemic stroke.
Components of primary composite endpoints separately. | 12 month after the inclusion of the last patient
  Cardiovascular events are: cardiovascular death, non-fatal AMI, non-fatal stroke, hospital admission for heart failure, and new hospitalization for unstable angina or TIA.
Number of re-vascularization procedures. | 12 month after the inclusion of the last patient
  Revascularisation procedures, including PCI, CABG, peripheral arterial revascularisation and intra-cerebral stent insertion
All-cause mortality. | 12 month after the inclusion of the last patient
  All-cause mortality.
New onset of ECG-confirmed atrial fibrillation or other arrhythmias. | 12 month after the inclusion of the last patient
  ECGs were performed at baseline and during the follow-up period; ECG and medical records were collected tovconfirm a hospitalization for atrial fibrillation event
Newly diagnosed diabetes mellitus, according to standard definitions. | 12 month after the inclusion of the last patient
  Newly diagnosed diabetes mellitus, according to standard definitions
Epworth Sleepiness Scale (ESS) and Test EuroQol (EQ-5D). | 12 month after the inclusion of the last patient
  OSA symptoms: Epworth Sleepiness Scale (ESS). Quality of life: Test EuroQol (EQ-5D).
Severity and phenotype of patients with OSA and clinical outcomes of ACS. | 12 month after the inclusion of the last patient
  To establish the relationship between the severity and phenotype of patients with OSA and clinical outcomes of ACS.
CPAP compliance and CV events incidence. | 12 month after the inclusion of the last patient
  To establish the relationship between CPAP compliance and CV events incidence.
Biological risk markers related to mechanisms involved in cardiovascular complications in these patients. | 12 month after the inclusion of the last patient
  To identify biological risk markers that allow us to establish the most important mechanisms involved in cardiovascular complications in these patients.
Cost-effectiveness analysis (Qualys) of the diagnosis and CPAP treatment of patients with ACS who have obstructive sleep apnea. | 12 month after the inclusion of the last patient
  Cost-effectiveness analysis (Qualys) of the diagnosis and CPAP treatment of patients with ACS who have obstructive sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbe, MD, Principal Investigator — Spanish Respiratory Sociey
Locations (1):
- Spanish Respiratory Society, Barcelona, Spain

REFERENCES:
- [Derived] Sanchez-de-la-Torre M, Gracia-Lavedan E, Benitez ID, Sanchez-de-la-Torre A, Moncusi-Moix A, Torres G, Loffler K, Woodman R, Adams R, Labarca G, Dreyse J, Eulenburg C, Thunstrom E, Glantz H, Peker Y, Anderson C, McEvoy D, Barbe F. Adherence to CPAP Treatment and the Risk of Recurrent Cardiovascular Events: A Meta-Analysis. JAMA. 2023 Oct 3;330(13):1255-1265. doi: 10.1001/jama.2023.17465. PMID 37787793
- [Derived] Pinilla L, Esmaeili N, Labarca G, Martinez-Garcia MA, Torres G, Gracia-Lavedan E, Minguez O, Martinez D, Abad J, Masdeu MJ, Mediano O, Munoz C, Cabriada V, Duran-Cantolla J, Mayos M, Coloma R, Montserrat JM, de la Pena M, Hu WH, Messineo L, Sehhati M, Wellman A, Redline S, Sands S, Barbe F, Sanchez-de-la-Torre M, Azarbarzin A. Hypoxic burden to guide CPAP treatment allocation in patients with obstructive sleep apnoea: a post hoc study of the ISAACC trial. Eur Respir J. 2023 Dec 7;62(6):2300828. doi: 10.1183/13993003.00828-2023. Print 2023 Dec. PMID 37734857
- [Derived] Sanchez-de-la-Torre M, Gracia-Lavedan E, Benitez ID, Zapater A, Torres G, Sanchez-de-la-Torre A, Aldoma A, de Batlle J, Targa A, Abad J, Duran-Cantolla J, Urrutia A, Mediano O, Masdeu MJ, Ordax-Carbajo E, Masa JF, De la Pena M, Mayos M, Coloma R, Montserrat JM, Chiner E, Minguez O, Pascual L, Cortijo A, Martinez D, Dalmases M, Lee CH, McEvoy RD, Barbe F; Spanish Sleep Network. Long-Term Effect of Obstructive Sleep Apnea and Continuous Positive Airway Pressure Treatment on Blood Pressure in Patients with Acute Coronary Syndrome: A Clinical Trial. Ann Am Thorac Soc. 2022 Oct;19(10):1750-1759. doi: 10.1513/AnnalsATS.202203-260OC. PMID 35442180
- [Derived] Reynor A, McArdle N, Shenoy B, Dhaliwal SS, Rea SC, Walsh J, Eastwood PR, Maddison K, Hillman DR, Ling I, Keenan BT, Maislin G, Magalang U, Pack AI, Mazzotti DR, Lee CH, Singh B. Continuous positive airway pressure and adverse cardiovascular events in obstructive sleep apnea: are participants of randomized trials representative of sleep clinic patients? Sleep. 2022 Apr 11;45(4):zsab264. doi: 10.1093/sleep/zsab264. PMID 34739082
- [Derived] Sanchez-de-la-Torre M, Sanchez-de-la-Torre A, Bertran S, Abad J, Duran-Cantolla J, Cabriada V, Mediano O, Masdeu MJ, Alonso ML, Masa JF, Barcelo A, de la Pena M, Mayos M, Coloma R, Montserrat JM, Chiner E, Perello S, Rubinos G, Minguez O, Pascual L, Cortijo A, Martinez D, Aldoma A, Dalmases M, McEvoy RD, Barbe F; Spanish Sleep Network. Effect of obstructive sleep apnoea and its treatment with continuous positive airway pressure on the prevalence of cardiovascular events in patients with acute coronary syndrome (ISAACC study): a randomised controlled trial. Lancet Respir Med. 2020 Apr;8(4):359-367. doi: 10.1016/S2213-2600(19)30271-1. Epub 2019 Dec 12. PMID 31839558
- [Derived] Bauca JM, Barcelo A, Fueyo L, Sanchis P, Pierola J, de la Pena M, Arque M, Gomez C, Morell-Garcia D, Sanchez-de-la-Torre A, Sanchez-de-la-Torre M, Abad J, Duran-Cantolla J, Mediano O, Masdeu MJ, Urrutia-Gajate A, Masa JF, Barbe F; Spanish Sleep Group. Biomarker panel in sleep apnea patients after an acute coronary event. Clin Biochem. 2019 Jun;68:24-29. doi: 10.1016/j.clinbiochem.2019.03.015. Epub 2019 Mar 28. PMID 30928393
- [Derived] Bauca JM, Yanez A, Fueyo L, de la Pena M, Pierola J, Sanchez-de-la-Torre A, Mediano O, Cabriada-Nuno V, Masdeu MJ, Teran-Santos J, Duran-Cantolla J, Masa JF, Abad J, Sanchez-de-la-Torre M, Barbe F, Barcelo A; Spanish Sleep Network. Cell Death Biomarkers and Obstructive Sleep Apnea: Implications in the Acute Coronary Syndrome. Sleep. 2017 May 1;40(5). doi: 10.1093/sleep/zsx049. PMID 28419383
- [Derived] Barcelo A, Bauca JM, Yanez A, Fueyo L, Gomez C, de la Pena M, Pierola J, Rodriguez A, Sanchez-de-la-Torre M, Abad J, Mediano O, Amilibia J, Masdeu MJ, Teran J, Montserrat JM, Mayos M, Sanchez-de-la-Torre A, Barbe F; Spanish Sleep Group. Impact of Obstructive Sleep Apnea on the Levels of Placental Growth Factor (PlGF) and Their Value for Predicting Short-Term Adverse Outcomes in Patients with Acute Coronary Syndrome. PLoS One. 2016 Mar 1;11(3):e0147686. doi: 10.1371/journal.pone.0147686. eCollection 2016. PMID 26930634
- [Derived] Torres G, Sanchez-de-la-Torre M, Barbe F. Relationship Between OSA and Hypertension. Chest. 2015 Sep;148(3):824-832. doi: 10.1378/chest.15-0136. PMID 25879807
- [Derived] Barbe F, Sanchez-de-la-Torre A, Abad J, Duran-Cantolla J, Mediano O, Amilibia J, Masdeu MJ, Flores M, Barcelo A, de la Pena M, Aldoma A, Worner F, Valls J, Castella G, Sanchez-de-la-Torre M; Spanish Sleep Network. Effect of obstructive sleep apnoea on severity and short-term prognosis of acute coronary syndrome. Eur Respir J. 2015 Feb;45(2):419-27. doi: 10.1183/09031936.00071714. Epub 2015 Jan 8. PMID 25573410
- [Derived] Esquinas C, Sanchez-de-la Torre M, Aldoma A, Flores M, Martinez M, Barcelo A, Barbe F; Spanish Sleep Network. Rationale and methodology of the impact of continuous positive airway pressure on patients with ACS and nonsleepy OSA: the ISAACC Trial. Clin Cardiol. 2013 Sep;36(9):495-501. doi: 10.1002/clc.22166. Epub 2013 Jul 10. PMID 23843147